CLINICAL TRIAL: NCT01460979
Title: Activity, Tolerability, Safety of Temsirolimus in Women With Ovarian Cancer Who Progressed During Previous Platinum Chemotherapy or Within 6 Months After Therapy or Advanced Endometrial Carcinoma
Brief Title: Efficacy,Tolerability,Safety of Temsirolimus in Women With Platinum-refractory Ovarian Carcinoma or Advanced Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-GYN 8
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Genital Diseases, Female; Ovarian Diseases; Ovarian Neoplasms; Endometrial Neoplasms
Keywords: Ovarian Cancer; Endometrial Carcinoma; Temsirolimus
MeSH Terms: conditions — Genital Diseases, Female; Ovarian Diseases; Ovarian Neoplasms; Endometrial Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental)
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — 25mg weekly intravenous until progression

SUMMARY:
The purpose of this study is to determine the activity, tolerability and safety of Temsirolimus in women with ovarian cancer who progressed during the previous platinum chemotherapy alternatively within 6 months from completion of therapy or advanced endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Before performance of study specific actions or assessment the patient has to be informed, has signed the written consent and is willing to follow the requirements concerning treatment and follow-up.Comment: Procedures which are according to common clinical routine and having been performed before having given written informed consent may be used for the purpose of screening procedures or initial medical assessment as long as these procedures follow the protocol.
* Required: negative pregnancy test in fertile women

Stratum A - Ovarian Cancer:

* Histologically confirmed Ovarian Cancer
* Platin-refractory relapsed disease: progression within a platin-based chemotherapy or within 6 months after completion of a platin-based chemotherapy
* Prior treatment with a taxane-based scheme
* minimum of one measurable or non-measurable tumor lesion(according to RECIST 1.1 criteria)
* Not more than 2 previous chemotherapies or cytostatic therapies (i.e. monoclonal antibodies, cytokines, signal transduction inhibitors)

Stratum B - Endometrian Cancer:

* Histologically confirmed Endometrian Cancer
* Advanced (International Federation of Gynaecology and Obstetrics (FIGO) III or IV) or relapsed diseases not amenable to potentially curative treatment with local surgery and/or radiation therapy
* Prior endocrine therapy is allowed
* Prior adjuvant chemotherapy is allowed
* Minimum of one measurable or non-measurable tumor lesion(according to RECIST 1.1 criteria)

Exclusion Criteria:

* ECOG > 2
* Prior therapy with mammalian target of rapamycin (mTOR) -Inhibitor
* Cytostatic therapy (i.e. monoclonal antibodies, cytokines, signal transduction inhibitors), cytotoxical chemotherapy or endocrine therapy or radiation at the same time
* Current or recent treatment with another study drug and/or participation in another clinical study within 28 days prior to first dose of study treatment
* Chemotherapy or cytostatic therapy (i.e. monoclonal antibodies, cytokines, signal transduction inhibitors) or radiation within 28 days prior to start of study treatment
* Known or supposed hypersensitivity compared to study medication
* Acute or chronical infection
* Second malignancy which influences the prognosis of the patient
* Inadequate renal function (Creatinin > 1.5 x Upper Limit of Normal (ULN))
* Inadequate liver function (aspartate transaminase (AST), alanine transaminase (ALT), gamma-Glutamyl transpeptidase (GGT) > 2.5 x ULN or > 5.0 x ULN in the presence of liver metastasis; Bilirubin > 1.5 x ULN)
* Platelets < 100.000 /μl; Absolute Neutrophil Count (ANC) < 1.500 /μl
* Cachectic patients with weight < 45kg
* Patients who need parenteral nutrition
* Patients with ileus within the last 28 days
* One of the following diseases within 12 months prior to first study treatment: myocardial infarction, severe/unstable angina, bypass surgery of the coronar- or peripheral vessels, symptomatic heart insufficiency, cerebrovascular insult, transient ischemic attack (TIA), pulmonary embolism, deep venous thrombosis, other thromboembolic events
* Current treatment with Cytochrome P450 3A4 (CYP3A4) -Inhibitors (i.e. protease inhibitors, antimycotics, calcium channel blocker, macrolide antibiotics, Cimetidine) or -inductors (i.e. Carbamazepin, Phenobarbital, Phenytoin, Rifampicin, amber)
* Uncontrolled hypertension (> 150/100 mmHg despite optimal medicinal treatment)
* Current cardiac arrhythmias (Common Terminology Criteria for Adverse Events of National Cancer Institute (NCI CTCAE) grade ≥ 2), atrial fibrillation, prolongation of QTc > 470 msec
* Left ventricular ejection fraction (LVEF) ≤ 50% defined by echocardiogram
* NCI CTCAE grade 3 hemorrhage within 4 weeks prior to beginning of treatment
* Symptoms which indicate brain metastases, spinal cord compression or give new indications for brain- or leptomeningeal metastases
* Human immunodeficiency virus (HIV) positive or manifested Acquired Immune Deficiency Syndrome (AIDS-disease)
* Patients with other severe diseases who represent an inadequate risk for study participation

Applicable only for patients with no hysterectomy and/or bilateral adnexectomy prior to start of study.

* lactation
* potential fertile women without adequate contraception (potential fertile women must use one of the following adequate contraception: complete abstinence, intrauterine spiral or another method with a failure quote < 1% per year)
* life expectancy < 3 months
* neurological or psychiatric diseases or drugs or alcohol abuse which suppose no adequate comprehension and consequently no effective consent to study participation or no acceptable compliance during the study
* predictable problems with the compliance to appointments for examinations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
progression-free survival | after 4 months for ovarian cancer and 6 months for endometrial carcinoma after study entry

SECONDARY OUTCOMES:
rate and duration of stable diseases according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 and Gynecologic Cancer Intergroup (GCIG)-criteria for ovarian cancer | every 8 weeks until progression
progression-free survival according to RECIST 1.1 and cancer antigen 125 (CA 125) (for ovarian cancer) (biological progression-free survival (PFSbio)) | every 8 weeks until progression
overall survival | weekly until progression; thereafter every 8 weeks
safety and toxicity, i.e. type, frequency, severity and duration of adverse reactions | weekly until progression; thereafter every 8 weeks
quality of life according to European Organisation for Research and Treatment of Cancer (EORTC) questionaires "QLQ C30", "QLQ OV28" and "QLQ-EN24" | every 8 weeks
rate and duration of stable diseases according to RECIST-criteria for endometrial cancer | every 8 weeks until progression

CONTACTS AND LOCATIONS:
Overall Officials: Günter Emons, Professor, Study Chair — AGO Study Group (Study Group of the Arbeitsgemeinschaft Gynaekologische Onkologie)
Locations (18):
- Germany (18):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universität Erlangen-Nürnberg, Erlangen, Bavaria
  - Klinikum rechts der Isar der Technischen Universität, München, Bavaria
  - GYNAEKOLOGICUM Bremen, Bremen, City state Bremen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Hesse
  - Universitätsklinikum Gießen-Marburg, Standort Marburg, Marburg, Hesse
  - Klinikum Offenbach, Offenbach, Hesse
  - Klinikum Göttingen, Georg-August-Universität, Göttingen, Lower Saxony
  - Gynäkologisch-onkologische Praxis, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Greifswald der Ernst-Moritz-Arndt-Universität, Greifswald, Mecklenburg-Vorpommern
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Kliniken Essen Mitte, Evang. Huyssens Stiftung/Knappschaft GmbH, Essen, North Rhine-Westphalia
  - Städt. Klinikum Solingen gGmbH, Solingen, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Charité, Campus Virchow Klinikum, Berlin, State of Berlin

REFERENCES:
- See also: Final publication — http://www.ncbi.nlm.nih.gov/pubmed/26731724